CLINICAL TRIAL: NCT03578029
Title: A Randomized,Single-Blind, Placebo-controlled, Self-matched Pairing, Independent Evaluated Study to Evaluate the Efficacy and Safety of RGN-137 Topical Gel in Subjects With Junctional and Dystrophic Epidermolysis Bullosa (CELEB)
Brief Title: Evaluation of the Safety and Efficacy Study of RGN-137 Topical Gel for Junctional and Dystrophic Epidermolysis Bullosa
Acronym: CELEB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Lenus Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGN-137-EB-202
Record Dates: First submitted 2018-06-14; First posted 2018-07-05 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Junctional Epidermolysis Bullosa; Dystrophic Epidermolysis Bullosa
Keywords: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa, Junctional; Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RGN-137 (Experimental): It is formulated as a gel for topical administration.
  Interventions: Drug: RGN-137
- Placebo (Placebo Comparator): It is composed of the same excipients as RGN-137 formulation without the active ingredient.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RGN-137 — It will be applied topically to the appropriate wound once a day for up to 84 days.
  Other Names: Dermal Topical Gel
  Arms: RGN-137
Drug: Placebo — It will be applied topically to the appropriate wound once a day for up to 84 days.
  Other Names: Vehicle Control
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the efficacy and safety of RGN-137 topical gel with that of placebo gel for treatment of junctional epidermolysis bullosa (JEB) or dystrophic epidermolysis bullosa (DEB).

DETAILED DESCRIPTION:
RGN-137 will be evaluated for efficacy and safety compared to a Placebo. A matched-pair design will be used to evaluate RGN-137 treatment versus placebo for treatment of 15 subjects with JEB or DEB. Eligible subject must have 1 set of matched-pair wound. The investigator will assign pair of index wounds, each wound with an area between 5cm2 and 50cm2, inclusive, for the eligible subject on Day 1, and for each pair, one wound will be randomized to receive RGN-137 gel and the other to receive Placebo gel. Subjects and independent evaluator will be blinded to the treatment assignments for each wound.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and at least 4 years old with a diagnosis of DEB or JEB
* Patients and their parents or guardians must be willing and able to provide written informed consent/assent
* Presence of 1 pair of stable index wounds within the specified size range at study

  1. Index wounds must have a surface area between 5 cm2 and 50 cm2, inclusive at the screening visit
  2. The index wounds selected as pairing must be relatively matched in terms of size and location
* Women of childbearing potential must have a negative pregnancy test prior to randomization
* Sexually active subjects must agree to use medically accepted methods of contraception during the study

Exclusion Criteria:

* Have any clinical evidence of local infection of the index lesion
* Use of prior or concomitant medication (Any investigational drug within 30 days, Immunotherapy or cytotoxic chemotherapy within 60 days, Systemic steroidal therapy within 30 days, and topical steroidal therapy within 14 days)
* History of sensitivity to any component of the treatment
* Neurological, cardiovascular, respiratory, hepatic, renal, or metabolic disease likely to interfere with the subject's participation in or completion of the study (At the discretion of investigator, participants with cardiomyopathy can participate)
* Current or former malignancy, including a history of squamous cell carcinomas
* Arterial or venous disorder resulting in ulcerated wounds
* Uncontrolled diabetes mellitus
* Pregnancy or breastfeeding during the study
* Girls or women who have had menarche but have not completed menopause
* Any condition or situation likely to cause the subject to be unable or unwilling to participate in the study procedures

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Time to achieving 50% reduction in area of each index wound from Day 1 up to Day 84. | up to Day 84
  This primary endpoint will the time to achieving 50% reduction in area of each index wound from Day 1 up to Day 84, defined as date of the first study visit on which 50% reduction in index wound area is achieved minus date of Day 1 visit.

SECONDARY OUTCOMES:
Time to achieving 50%, 75%, and 100% (with drainage or without drainage) reduction in area of each index wound from Day 1 up to Day 84. | up to Day 84
  This secondary endpoint will the time to achieving 50%, 75%, and 100% reduction in area of each index wound from Day 1 up to Day 84, defined as date of the first study visit on which 50% reduction in index wound area is achieved minus date of Day 1 visit.
Incidence of 50%, 75%, and 100% reduction and complete re-epithelialization without drainage in area of each index wound at the scheduled visits. | up to Day 84
  This secondary endpoint will be summarized by treatment using frequency counts and percentages.
Change from Baseline and percent change from Baseline in surface area of each index wound at the scheduled visits. | up to Day 84
  This secondary endpoint will be computed for each treatment group as well as for treatment difference at each visit.

OTHER OUTCOMES:
Index wound characteristics at the scheduled visits. | up to Day 84
  (inflammation/erythema, induration, crusting, exudate, cellulitis, and other abnormalities)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northwestern University, Evanston, Illinois
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Dermatology and Laser Specialists, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No